CLINICAL TRIAL: NCT00119132
Title: A Study Of Impact Of Intermittent Preventive Treatment In Children With Amodiaquine Plus Artesunate Versus Sulphadoxine-Pyrimethamine On Hemoglobin Levels And Malaria Morbidity In Hohoe District Of Ghana
Brief Title: Effectiveness of Intermittent Preventive Treatment for Malaria in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: INDEPTH Network (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ITCR5098
Record Dates: First submitted 2005-07-04; First posted 2005-07-13 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: intermittent preventive treatment; effectiveness; malaria
MeSH Terms: conditions — Malaria | interventions — amodiaquine, artesunate drug combination; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: artesunate-amodiaquine
Drug: sulphadoxine-pyrimethamine

SUMMARY:
Intermittent preventive treatment for malaria in children (IPTc) is a promising new approach to malaria control. Preliminary studies of IPTc in Senegal and Mali indicate that this approach can be very effective. Although the results of these studies suggest that IPTc with sulphadoxine-pyrimethamine (SP) plus artesunate (AS) or SP alone is an efficacious and safe intervention for reducing the burden of malaria and anaemia in children in high transmission areas with short transmission periods, there is no data from areas with long transmission periods. This study aims to evaluate the effectiveness of IPTc in reducing anaemia and malaria in an area with up to 6 months of transmission in Ghana. Two thousand two hundred forty children aged 3-59 months will be randomly allocated to four groups (560 per arm) to receive amodiaquine plus artesunate (AQ+AS), given at two different intervals (monthly or bimonthly), SP or placebo. The children will also be followed to determine if there is any rebound in the incidence of severe malaria and anaemia in the year following IPTc.

DETAILED DESCRIPTION:
Background:

In high transmission areas, where a major proportion of deaths and severe morbidity from malaria occurs during the first year of life, intermittent preventive treatment for infants (IPTi) could make a major contribution to reducing the burden of malaria as a whole. However, in many areas in Africa, where mortality and morbidity from malaria in children under five years of age is very high and the burden of malaria is not predominantly in infants, IPTi, even if highly effective, would have only a limited impact on the overall burden of malaria in children.

Few community trials have evaluated the effect of IPTc in the prevention of malaria. Dicko and his colleagues in Mali, an area of seasonal malaria transmission gave two doses of SP to children aged 6 months to 9 years at an interval of two months and found a protective efficacy of 40% against clinical attacks of malaria among children in the intervention group compared to the placebo group. Recent work in Niakhar, Senegal has assessed IPTc in an area of intense but short seasonal malaria transmission. The study used a combination of SP plus one dose of AS, which was given every month for three months during the rainy season which lasted for only four months. This study showed that IPTc using AS+SP was well tolerated without any drug-attributable adverse events and that IPTc can reduce the incidence of clinical malaria by 86%. Although these results suggest that IPTc with SP+one dose of AS is an efficacious and safe intervention for reducing the burden of malaria and anaemia in children, there is no data on the effectiveness of IPTc in areas with prolonged transmission seasons and on the use of other forms of combination therapy in IPTc.

Study overview:

The study aims to determine the optimum drug schedule for IPTc in an area of prolonged seasonal malaria transmission in Ghana. The main study will compare the effectiveness of IPTC using SP, monthly AQ+AS or bimonthly AQ+AS. In order to facilitate the interpretation of the results of this trial, two ancillary studies will be done. The first will be a conventional in vivo drug efficacy study of SP and AQ+AS in children with clinical malaria to ensure the efficacy of the drugs used in the IPTc trial within the study area. The second subsidiary study will be an investigation of whether or not administration of IPTc over one malaria transmission season is followed by an increase in the incidence of malaria or anaemia during the following malaria transmission season.

Study Objectives:

1. To investigate whether IPTc using monthly or bimonthly AQ+AS or SP can improve mean Hb level and decrease anaemia and malaria morbidity in young children in an area of intense and prolonged seasonal malaria transmission.
2. To compare the incidence of severe malaria among children aged 3-59 months using the three treatment regimens.

Study area:

The study will be carried out in Hohoe district, Ghana. The major rainy season lasts from April to July and the minor one from September to November. The rest of the year is relatively dry. Malaria is the most common disease in this area. For the past four years malaria has accounted for 32% of the out patient attendances out of which 45% were children under five years. Twenty five percent (25%) of malaria cases required inpatient care and 37% of the cases were children under five years and 57% of them reported with anaemia. The peak of OPD malaria and anaemia cases occurs between June and October.

Study procedures:

A cross-sectional survey will be carried out after informed consent has been obtained from the guardians of all children aged between 3 to 59 months in the selected villages. Information will be collected on the background of the child and guardian, hypersensitivity to the study drugs and bednet use. Anthropometric indices will be measured.

Drugs will be administered to the study children every month from May to October. Field workers and coordinators will visit the participants once a week from May to October. Parents and guardians will be strongly advised to come directly to a health centre if their child develops any symptoms or signs of illness between the field workers' weekly home-visits. Passive surveillance will be performed by six medical assistants and twelve nurses based in the health centres in the sub-districts within the district. Malaria clinical attacks will be documented and treatment for malaria and any other illness will be provided free of charge to study participants in all the health centres that are in the catchment area of the selected communities.

If the child has fever or any features suggestive of malaria, a finger prick blood sample will be collected for Hb and malaria parasite detection. Two slides will be prepared for each child. At the health centre, one slide will be examined on the same day for deciding on appropriate treatment. The second slide will be kept and sent to the central laboratory for reading to provide a definitive diagnosis. Those who have malaria will be treated with oral quinine 10mg/kg every 8 hours for 7days and will be followed on days 3 and 7 for outcome measurement.

At the end of the malaria transmission season, a cross-sectional survey will be undertaken involving all children who have remained in the study. Following administration of a short questionnaire, a finger prick blood sample will be obtained for preparation of a blood film and for determination of Hb. A filter paper sample will be collected for molecular studies.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3-59 months resident in the selected communities
* Children likely to be available for follow-up for 18 months
* Consent by parent/guardian of child

Exclusion Criteria:

* Chronic illness
* History of hypersensitivity to any of the study drugs

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2602 (Actual)
Dates: Start 2005-06; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Mean Hb at the end of the high transmission season.

SECONDARY OUTCOMES:
Incidence of moderate (Hb<8.0g/dl>5.0g/dl) and severe anaemia (Hb<5.0g/dl) during the period of the intervention
Incidence of severe and clinical malaria during the period of the intervention
Prevalence of anaemia at the post intervention survey
Prevalence of parasitaemia and gametocytemia at the post intervention survey
Prevalence of molecular markers of resistance to SP among children who have malaria at the post intervention survey

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kweku, MBChB, MPH, Principal Investigator — London School of Hygiene and Tropical Medicine; Daniel Chandramohan, MBBS, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Brian Greenwood, FRCP, FRS, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Ministry of Health, Hohoe district hospital, Hohoe, Volta Region, Ghana

REFERENCES:
- [Derived] Patouillard E, Conteh L, Webster J, Kweku M, Chandramohan D, Greenwood B. Coverage, adherence and costs of intermittent preventive treatment of malaria in children employing different delivery strategies in Jasikan, Ghana. PLoS One. 2011;6(11):e24871. doi: 10.1371/journal.pone.0024871. Epub 2011 Nov 3. PMID 22073137
- [Derived] Conteh L, Patouillard E, Kweku M, Legood R, Greenwood B, Chandramohan D. Cost effectiveness of seasonal intermittent preventive treatment using amodiaquine & artesunate or sulphadoxine-pyrimethamine in Ghanaian children. PLoS One. 2010 Aug 17;5(8):e12223. doi: 10.1371/journal.pone.0012223. PMID 20808923
- [Derived] Kweku M, Webster J, Adjuik M, Abudey S, Greenwood B, Chandramohan D. Options for the delivery of intermittent preventive treatment for malaria to children: a community randomised trial. PLoS One. 2009 Sep 30;4(9):e7256. doi: 10.1371/journal.pone.0007256. PMID 19789648
- [Derived] Kweku M, Liu D, Adjuik M, Binka F, Seidu M, Greenwood B, Chandramohan D. Seasonal intermittent preventive treatment for the prevention of anaemia and malaria in Ghanaian children: a randomized, placebo controlled trial. PLoS One. 2008;3(12):e4000. doi: 10.1371/journal.pone.0004000. Epub 2008 Dec 22. PMID 19098989